CLINICAL TRIAL: NCT02511431
Title: Treatment of Chronic Delta Hepatitis With Lonafarnib and Ritonavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150170; 15-DK-0170
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2017-02-23

CONDITIONS: Hepatitis D
Keywords: Delta Hepatitis; Hepatitis D; Liver Disease; Hepatitis D Virus; Chronic Hepatitis
MeSH Terms: conditions — Hepatitis D; Liver Diseases; Hepatitis, Chronic | interventions — lonafarnib; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Lonafarnib/Ritonavir at 50 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- Group 2 (Experimental): Lonafarnib/Ritonavir at 75 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- Group 3 (Experimental): Lonafarnib/Ritonavir at 100 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- Group 4 (Experimental): Placebo for 12 weeks then Lonafarnib/Ritonavir at 50 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir; Other: Placebo
- Group 5 (Experimental): Placebo for 12 weeks then Lonafarnib/Ritonavir at 75 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir; Other: Placebo
- Group 6 (Experimental): Placebo for 12 weeks then Lonafarnib/Ritonavir at 100 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Interventions: Drug: Lonafarnib; Drug: Ritonavir; Other: Placebo

INTERVENTIONS:
Drug: Lonafarnib — prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
Drug: Ritonavir — FDA approved drug for use of boosting other drugs. Will be used to boost Lonafarnib as they both use the same cytochrome P450 system. Will be administered at 100 mg daily.
Other: Placebo — Placebo
  Arms: Group 4; Group 5; Group 6

SUMMARY:
Background:

- Chronic hepatitis D is a liver disease caused by the hepatitis D virus (HDV). It can be severe and progressive. Most people with hepatitis D will develop scarring and damage to the liver. There is no FDA approved drug to treat chronic hepatitis D. Researchers want to know if the drugs lonafarnib and ritonavir can help people with chronic hepatitis D.

Objective:

- To find out if treatment of hepatitis D with lonafarnib and ritonavir is safe and effective.

Eligibility:

- People 18 years of age and older with chronic hepatitis D. They must not have HIV or other major illnesses.

Design:

* Participants will be screened with medical history, physical exams, and blood tests.
* Participants will have 24 weeks of treatment. They will then have 24 weeks of follow-up.
* Participants will be in 1 of 6 treatment groups. Those in each group will receive different doses of the study drugs. Some groups will start with placebo but will receive treatment after 3 months of placebo.
* Participants will also take drugs to treat hepatitis B.
* Participants will have many visits. These will include:
* One three-day stay at the Clinical Center
* Physical exams
* EKG: small sticky patches will be put on the chest, arms, and legs to trace heart rhythm
* Ultrasounds of the abdomen
* Urine and blood tests
* Stool samples
* Eye exams
* Evaluations by a reproductive endocrinologist (women) or urologist (men). Men may provide a sperm sample (optional).

DETAILED DESCRIPTION:
Chronic delta hepatitis is a serious form of chronic liver disease caused by infection with the hepatitis D virus (HDV), a small RNA virus that requires farnesylation of its major structural protein (HDV antigen) for replication. We propose to treat 21 adult patients with chronic delta hepatitis using the combination of the farnesyltransferase inhibitor (FTI) lonafarnib (LNF) and the protease inhibitor ritonavir (RTV). LNF has been shown to decrease serum quantitative HDV RNA in patients with chronic delta hepatitis infection, but dosing is limited by its side effects. RTV inhibits one of the cytochrome P-450 systems that metabolizes LNF leading to higher serum levels of LNF with minimal side effects. In this randomized, double-blinded, placebo-controlled study, there will be six groups of patients; Group 1(4 patients) will receive LNF/RTV 50/100 mg daily for 24 weeks, Group 2 (4 patients) will receive LNF/RTV 75/100mg daily for 24 weeks, Group 3 (4 patients) will receive LNF/RTV 100/100mg daily for 24 weeks, Group 4, 5 and 6 (3 patients for each group) will initially receive placebo for 12 weeks followed by either LNF/RTV 50/100 mg daily (3 patients) or LNF/RTV 75/100mg daily (3 patients) or LNF/RTV 100/100 mg daily (3 patients) for 12 weeks. After dosing, all patients will be monitored for 24 weeks off therapy. Nucleos(t)ide analogue therapy will be instituted during this study to prevent the possibility of hepatitis B virus reactivation/flare; Patients on pre-existing nucleos(t)ide analogues will be continued and patients not on pre-existing therapy will receive either entecavir or tenofovir for 48 weeks. Patients with quantifiable HDV RNA in serum and elevated aminotransferases will be enrolled. Before receiving therapy, patients will be evaluated for at least 3 visits with regular testing for HDV RNA quantitation and alanine aminotransferase (ALT) levels and will undergo Clinical Center admission for medical evaluation, timed blood draws and to start therapy. At each clinic visit, patients will be questioned about side effects, symptoms and quality of life, undergo focused physical examination, and have blood drawn for complete blood counts, HDV RNA, and routine liver tests (including ALT, aspartate aminotransferase , alkaline phosphatase, direct and total bilirubin, and albumin). At the end of the treatment, patients will undergo repeat physical examination, assessment of symptoms (using a symptom scale questionnaire), complete blood counts, routine liver tests, and hepatitis B and D viral markers. The primary therapeutic endpoint will be a decline of HDV RNA viral titer of 2 logs at the end of therapy. The primary safety endpoint will be the ability to tolerate the drugs at the prescribed dose for the full course of therapy. Several secondary endpoints will be measured, including side effects, ALT levels, maintained virological response, undetectable HDV RNA in the serum, loss of HBsAg and symptoms. Therapy will be stopped for intolerance to lonafarnib and/or ritonavir (which will be carefully defined). This clinical trial is designed as a phase 2a study assessing the antiviral activity, safety and tolerance of three different doses of lonafarnib and ritonavir.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years or above, male or female.
  2. Serum alanine or aspartate aminotransferase (ALT or AST) activities above the upper limit of normal (ALT greater than or equal to 20 or AST greater than or equal to 20 U/L in females and ALT greater than or equal to 30 or AST greater than or equal to 30 U/L in males) on an average of three determinations taken during the previous 6 months at the NIH clinical center. The mean of the three determinations will be defined as baseline levels.
  3. Presence of anti-HDV in serum.
  4. Presence of quantifiable HDV RNA in serum.

EXCLUSION CRITERIA:

1. Decompensated liver disease, defined by bilirubin >4mg/dL, albumin <3.0 gm/dL, prothrombin time >2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Laboratory abnormalities that are not thought to be due to liver disease may not necessarily require exclusion. Patients with ALT levels greater than 1000 U/L (>25 times ULN) will not be enrolled but may be followed until three determinations are below this level.
2. Pregnancy, active breast-feeding, or inability to practice adequate contraception, in women of childbearing potential or in spouses of such women. Adequate contraception is defined as vasectomy in men, tubal ligation in women, or use of two barrier methods such as condoms and spermicide combination, birth control pills, an intrauterine device, Depo-Provera, or Norplant. In total, the participant and their partner must utilize two forms of contraception and one method must include a barrier method.
3. Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR <50 ml/min), organ transplantation, serious psychiatric disease or depression (only if felt to be at high risk by the NIH psychiatric consultation service), and active coronary artery disease.
4. Systemic immunosuppressive therapy within the previous 2 months.
5. Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, alcoholic liver disease, nonalcoholic steatohepatitis (but not steatosis), hemochromatosis, or alpha-1-antitrypsin deficiency).
6. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.
7. Evidence of hepatocellular carcinoma.
8. Evidence of concurrent hepatitis C infection with positive serum hepatitis c virus (HCV) RNA.
9. Any experimental therapy or pegylated interferon therapy within 6 months prior to enrollment.
10. Diagnosis of malignancy in the five years prior to the enrollment with exception granted to superficial dermatologic malignancies.
11. Evidence of HIV co-infection; HIV 1/2 viral RNA or antigen on serum testing.
12. Concurrent usage of statins as these drugs inhibits mevalonate synthesis, which reduces protein prenylation.
13. Concurrent usage of moderate and strong cytochrome p450, family 3, subfamily A (CYP3A) inhibitors and inducers.
14. Use of any prescription, nonprescription or natural medicine (herbal) medications unless the use of medication is medically necessary with appropriate monitoring.
15. Concurrent usage of alpha 1 adrenoreceptor antagonist, antiarrhythmic, pimozide, sildenafil, sedative and hypnotics, ergot and St. John s Wort due to possible effect of ritonavir on hepatic metabolism of these drugs resulting in potentially life threatening side effects.
16. Clinically significant baseline EKG abnormalities.
17. Uncontrolled elevated triglycerides.
18. History of pancreatitis as a result of hypertriglyceridemia.
19. Inability to understand or sign informed consent.
20. Any other condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-29; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kefalakes H, Koh C, Sidney J, Amanakis G, Sette A, Heller T, Rehermann B. Hepatitis D Virus-Specific CD8+ T Cells Have a Memory-Like Phenotype Associated With Viral Immune Escape in Patients With Chronic Hepatitis D Virus Infection. Gastroenterology. 2019 May;156(6):1805-1819.e9. doi: 10.1053/j.gastro.2019.01.035. Epub 2019 Jan 18. PMID 30664876
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0170.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment number in the Protocol Section (22) conflicts with the number of participants started (21). One enrolled patient declined participation prior to randomization.
Groups:
- 50mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 50 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same cytochrome p450 (CYP) system. Will be administered at 100 mg daily.
- 75mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 75 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
- 100mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 100 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
- Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir: Placebo for 12 weeks then Lonafarnib/Ritonavir at 50 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
  Placebo: Placebo
- Placebo Then 75mg/100mg Lonafarnib/Ritonavir: Placebo for 12 weeks then Lonafarnib/Ritonavir at 75 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
  Placebo: Placebo
- Placebo Then 100mg/100mg Lonafarnib/Ritonavir: Placebo for 12 weeks then Lonafarnib/Ritonavir at 100 mg/100 mg daily for 12 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
  Placebo: Placebo
Period: Treatment
Arm/Group | 50mg/100mg Lonafarnib/Ritonavir | 75mg/100mg Lonafarnib/Ritonavir | 100mg/100mg Lonafarnib/Ritonavir | Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir | Placebo Then 75mg/100mg Lonafarnib/Ritonavir | Placebo Then 100mg/100mg Lonafarnib/Ritonavir
Started | 4 | 4 | 4 | 3 | 3 | 3
Completed | 4 | 4 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1
Period: Post-treatment Follow-up
Arm/Group | 50mg/100mg Lonafarnib/Ritonavir | 75mg/100mg Lonafarnib/Ritonavir | 100mg/100mg Lonafarnib/Ritonavir | Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir | Placebo Then 75mg/100mg Lonafarnib/Ritonavir | Placebo Then 100mg/100mg Lonafarnib/Ritonavir
Started | 4 | 4 | 3 | 3 | 3 | 2
Completed | 4 | 4 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 50mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 50 mg/100 mg daily for 24 weeks followed by 24 weeks of off therapy follow-up.
  Lonafarnib: prenylation inhibitor to be administered daily at doses of 50 mg, 75 mg or 100 mg.
  Ritonavir: FDA approved drug for use of boosting other drugs. Will be used to boost ritonavir as they both use the same CYP system. Will be administered at 100 mg daily.
- Total: Total of all reporting groups
Arm/Group | 50mg/100mg Lonafarnib/Ritonavir | 75mg/100mg Lonafarnib/Ritonavir | 100mg/100mg Lonafarnib/Ritonavir | Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir | Placebo Then 75mg/100mg Lonafarnib/Ritonavir | Placebo Then 100mg/100mg Lonafarnib/Ritonavir | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 21
Age, Continuous [Median (Full Range); unit: years] | 48 [34 to 66] | 43.5 [22 to 53] | 40.5 [31 to 45] | 39 [30 to 53] | 52 [47 to 54] | 45 [33 to 47] | 45 [22 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 2 | 2 | 0 | 8
  Male | 2 | 2 | 4 | 1 | 1 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 1 | 2 | 1 | 1 | 9
  Black | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Multiple | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 2 | 2 | 1 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decline of Hepatitis Delta Virus (HDV) RNA Quantitative Measurements of >2 Logs From Baseline at 12 Weeks of Treatment
Description: The number of participants who experienced a > 2 log IU/mL decline in serum HDV RNA at 12 weeks of treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg/100mg Lonafarnib/Ritonavir | 75mg/100mg Lonafarnib/Ritonavir | 100mg/100mg Lonafarnib/Ritonavir | Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir | Placebo Then 75mg/100mg Lonafarnib/Ritonavir | Placebo Then 100mg/100mg Lonafarnib/Ritonavir
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 2
Participants | 1 | 1 | 1 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Decline of HDV RNA Quantitative Measurement of > 2 Logs From Baseline at 24 Weeks of Treatment
Description: The number of participants who experienced a > 2 log IU/mL decline in serum HDV RNA levels at 24 weeks of treatment
Time Frame: 24 weeks
Population: This outcome is for decline in serum HDV RNA levels over 24 weeks of treatment. Arms 4, 5 and 6 had only 12 weeks of treatment and so are not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg/100mg Lonafarnib/Ritonavir | 75mg/100mg Lonafarnib/Ritonavir | 100mg/100mg Lonafarnib/Ritonavir | Placebo Then 50 mg/100 mg Lonafarnib/Ritonavir | Placebo Then 75mg/100mg Lonafarnib/Ritonavir | Placebo Then 100mg/100mg Lonafarnib/Ritonavir
Number analyzed (Participants) | 4 | 4 | 3 | 0 | 0 | 0
Participants | 1 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For the 12 patients in arms 1, 2 and 3 (24 weeks of treatment), adverse event data were collected over the 24 weeks of treatment and are reported per arm. For patients in arms 4, 5 and 6 (12 weeks placebo then 12 weeks active treatment), adverse event data for the placebo portion of the study were collected over the 12 weeks of placebo administration (reported in aggregate) and the 12 weeks of active treatment (reported per arm).
Groups:
- 24 Weeks of 50mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 50 mg/100 mg daily for 24 weeks.
- 24 Weeks of 75mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 75 mg/100 mg daily for 24 weeks.
- 24 Weeks of 100mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 100 mg/100 mg daily for 24 weeks.
- 12 Weeks of Placebo: Placebo for first 12 weeks.
- 12 Weeks of 50 mg/100 mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 50 mg/100 mg daily for second 12 weeks.
- 12 Weeks of 75mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 75 mg/100 mg daily for second 12 weeks.
- 12 Weeks of 100mg/100mg Lonafarnib/Ritonavir: Lonafarnib/Ritonavir at 100 mg/100 mg daily for second 12 weeks.
Arm/Group | 24 Weeks of 50mg/100mg Lonafarnib/Ritonavir | 24 Weeks of 75mg/100mg Lonafarnib/Ritonavir | 24 Weeks of 100mg/100mg Lonafarnib/Ritonavir | 12 Weeks of Placebo | 12 Weeks of 50 mg/100 mg Lonafarnib/Ritonavir | 12 Weeks of 75mg/100mg Lonafarnib/Ritonavir | 12 Weeks of 100mg/100mg Lonafarnib/Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/9 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 0/4 | 0/9 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 3/4 | 8/9 | 3/3 | 3/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24 Weeks of 50mg/100mg Lonafarnib/Ritonavir (N=4) | 24 Weeks of 75mg/100mg Lonafarnib/Ritonavir (N=4) | 24 Weeks of 100mg/100mg Lonafarnib/Ritonavir (N=4) | 12 Weeks of Placebo (N=9) | 12 Weeks of 50 mg/100 mg Lonafarnib/Ritonavir (N=3) | 12 Weeks of 75mg/100mg Lonafarnib/Ritonavir (N=3) | 12 Weeks of 100mg/100mg Lonafarnib/Ritonavir (N=3)
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 24 Weeks of 50mg/100mg Lonafarnib/Ritonavir (N=4) | 24 Weeks of 75mg/100mg Lonafarnib/Ritonavir (N=4) | 24 Weeks of 100mg/100mg Lonafarnib/Ritonavir (N=4) | 12 Weeks of Placebo (N=9) | 12 Weeks of 50 mg/100 mg Lonafarnib/Ritonavir (N=3) | 12 Weeks of 75mg/100mg Lonafarnib/Ritonavir (N=3) | 12 Weeks of 100mg/100mg Lonafarnib/Ritonavir (N=3)
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 3 | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 3 | 4 | 2 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 5 | 1 | 2 | 1
Bloating (Gastrointestinal disorders) | 2 | 1 | 2 | 4 | 1 | 3 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 5 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT02511431/Prot_SAP_000.pdf